CLINICAL TRIAL: NCT06627218
Title: Liberal or Adhere to Recommendations for Prothrombin Complex Concentrate Management in Major Bleeding Following Trauma：A Multicenter Retrospective Study
Brief Title: Liberal or Adhere to Recommendations for PCC Management in Major Bleeding Following Trauma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0580
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-09

CONDITIONS: Traumatic Bleeding
Keywords: trauma; Major Bleeding
MeSH Terms: conditions — Wounds and Injuries | interventions — Factor IX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adhere to Recommendations for PCC Management (Experimental): Adhere to Recommendations for PCC Management in Major Bleeding Following Trauma
  Interventions: Drug: Prothrombin Complex Concentrate
- Liberal PCC Management (No Intervention): Liberal PCC Management in Major Bleeding Following Trauma

INTERVENTIONS:
Drug: Prothrombin Complex Concentrate — Adhere to Recommendations for PCC Management in Major Bleeding Following Trauma
  Other Names: test group
  Arms: Adhere to Recommendations for PCC Management

SUMMARY:
Severe post-traumatic bleeding remains a major challenge in trauma management . The effectiveness and safety of PCC in the treatment of major traumatic bleeding is controversial, and the indications for use are not clear. Studies on the status of PCC use and the efficacy evaluation of PCC adhere to recommendations are lacking.

DETAILED DESCRIPTION:
Post-traumatic severe bleeding and associated traumatic coagulopathy remains a challenge.

The use of prothrombin complex concentrate (PCC) is being explored in the management of on-going coagulopathy following trauma, with the cited purpose of boosting thrombin generation. Clinical data on the efficacy of PCC as part of a coagulation factor concentrate-based haemostatic strategy showed initial promising results in retrospective studies and meta-analysis.

Certainly, the utility of PCC was a residual question in the management of traumatic coagulopathy. Uncertainty remains on the indication of use.The 2019 guideline on management of major bleeding and coagulopathy following trauma suggest that PCC should be administered to the bleeding patient based on evidence of delayed coagulation initiation using VEM, provided that fibrinogen levels are normal. The recommendation Grade is 2C.Studies on the status of PCC use and the efficacy evaluation of PCC adhere to recommendations are lacking.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old or < 80 years old
2. Trauma treated in resuscitation unit/emergency room patient
3. Hospital admission within 24h after injury
4. Assessment of blood consumption (ABC) score ≥2 points.

Exclusion Criteria:

1. PCC was used before admission
2. Anticoagulant drugs (such as low molecular weight heparin, rivaroxaban, warfarin, etc.)
3. Previous venous thrombosis (VTE, Patients with a history of coronary artery stents within 3 months of pulmonary embolism and myocardial infarction)
4. Patients with traumatic cardiac arrest in hospital
5. Women during breastfeeding, pregnancy or pregnancy
6. Patients with hemophilia A and other blood system diseases, severe liver disease, cirrhosis and other coagulation dysfunction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
in-hospital mortality | 14 days
  in-hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: yongan xu, doctor, Study Chair — Department of Emergency medicine，Second Affiliated Hospital of Zhejiang University
Locations (1):
- Department of Emergency medicine, Second Affiliated Hospital, School of Medicine& Institute of Emergency medicine, Zhejiang University,, Hangzhou, Zhejiang, China